CLINICAL TRIAL: NCT00779077
Title: An Open, Observational, Non-Interventional Study of Inspiratory Flow Rates and Volumes in Subjects With Cystic Fibrosis Inhaling Via a Spirometer With the High Resistance RS01 Dry Powder Inhaler Device in Series
Brief Title: Cystic Fibrosis (CF) Flow Rates Study
Status: Completed | Type: Observational
Sponsor: Syntara (Industry)
Responsible Party: Dr Brett Charlton, Pharmaxis
Other Study IDs: DPM-OSM-403
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Cystic Fibrosis
Keywords: device characteristics
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cystic fibrosis: adults and children with cystic fibrosis

SUMMARY:
We wish to measure the inspiratory flow and volumes generated by the subjects inhaling from a spirometer with a high resistance dry powder inhaler in series in subjects with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* CF
* FEV1 ≥ 30% and < 90% predicted

Exclusion Criteria:

* Be considered "terminally ill" or listed for lung transplantation
* Have had a lung transplant
* Have had a significant episode of haemoptysis (>60 ml) in the three months prior to enrolment
* Have had a myocardial infarction in the three months prior to enrolment
* Have had a cerebral vascular accident in the three months prior to enrolment
* Have had major ocular surgery in the three months prior to enrolment
* Have had major abdominal, chest or brain surgery in the three months prior to enrolment
* Have a known cerebral, aortic or abdominal aneurysm
* Be breast feeding or pregnant
* Be using beta blockers
* Have unstable asthma

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CF 6yrs and above
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
inspiratory flow rates | single visit

SECONDARY OUTCOMES:
inspiratory volumes | single visit